CLINICAL TRIAL: NCT03487497
Title: Gait Analysis During Level and Uphill Walking After Lengthening Osteotomy of the Lateral Column
Acronym: CALCOT
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-00254
Record Dates: First submitted 2018-02-28; First posted 2018-04-04 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Osteotomy; Lengthening; Leg
Keywords: gait analysis; electromyography; strength test; walking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients who underwent lateral column lengthening osteotomy
  Interventions: Procedure: Lateral column lengthening osteotomy
- Healthy subjects: Healthy subjects without intervention

INTERVENTIONS:
Procedure: Lateral column lengthening osteotomy — Lengthening osteotomy of the lateral column of the foot
  Groups: Patients

SUMMARY:
A common surgical treatment for posterior tibial tendon dysfunction (and the resulting flat foot) is the correction through a calcaneal lengthening osteotomy of the lateral column (LLC). Clinical studies showed pain relief and functional improvements through different scores. However, according to clinical experience, some patients complain about a limited ankle dorsiflexion after LLC surgery. Several joints of the foot (talocrural, subtalar, talonavicular, calcaneocuboid) contribute to the overall range of motion in foot plantarflexion/dorsiflexion and pronation/supination. Changes in the range of motion in one joint can affect all the other joints. For instance, it was shown that a fusion of the talonavicular joint removes most of the residual hindfoot motion in plantarflexion/dorsiflexion and pronation/supination. Because the lengthening of the lateral column presumably decreases the mobility of the medial column and thus of the talonavicular joint, this surgery can influence the range of motion of the other joints, and hence contribute to the reported decreased ankle dorsiflexion motion.

Patients after LLC have less plantarflexion of the first metatarsal throughout stance of level walking and less inversion of the hindfoot during push-off compared to healthy subjects. Uphill walking requires more ankle plantarflexion and dorsiflexion than level walking. A limitation of the ankle joint mobility especially in dorsiflexion could therefore lead to additional or greater changes in gait patterns (hindfoot and forefoot kinematics) during uphill walking.

The primary objective is:

• To compare differences in hindfoot and forefoot kinematics between level and uphill treadmill walking in relation to passive range of motion

The secondary objectives are:

* To compare lower leg muscle activation during level and uphill treadmill walking between patients after LLC and healthy subjects
* To test the association between muscle strength, muscle activation patterns and hindfoot and forefoot kinematics during level and uphill walking and heel rise
* To relate clinical outcome of LLC surgery by functional scores to passive range of motion

DETAILED DESCRIPTION:
At the initial assessment, written informed consent will be obtained before participants will undergo a clinical exam (inspection and palpation of the foot, measurement of bilateral passive ankle range of motion). All participants will complete the Short Form (SF)36 and the Foot Function Index20 to obtain pain and functional scores (approximate duration: 30 minutes). Participants will be able to familiarize with treadmill walking at their preferred walking speed. Surface electrodes will be placed bilaterally over the tibialis anterior, gastrocnemius medialis and lateralis, soleus, and peroneus brevis. Isokinetic muscle strength in ankle plantarflexion/ dorsiflexion and inversion/eversion will be tested using the Biodex system 4 Pro (approximate duration: 45 minutes). Reflective surface markers will be placed bilaterally on anatomic landmarks according to the Plug In Gait model and a specific foot model. These markers are seen by 6 Vicon MX cameras. Participants will be asked to stand on the treadmill (h/p cosmos, Zebris), and data for a standing reference trial will be collected. Single-limb heel rise performance with each leg will be tested on the treadmill while kinematic, electromyography (EMG), and pressure data will be measured. Participants will then walk barefoot for 2 minutes at 0% slope while kinematic, EMG, and pressure data will be recorded. Subsequently, the treadmill incline will be increased to 15%, and data for 2 minutes walking at this slope will be recorded followed by three heel rises (approximate duration: 45 minutes). The estimated total time for each participant is 120 minutes.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* age < 70 years
* Patients:
* Unilateral surgery for posterior tibial tendon dysfunction by flexor digitorum longus transfer and lateral lengthening osteotomy of the calcaneus
* Minimum of 2 years postoperatively

Exclusion Criteria:

* Neuromuscular disorders affecting gait
* Cardiovascular disease
* Diabetes
* Pregnancy (if unknown, a pregnancy test (urine test) will be performed)
* Body mass index > 35 kg/m2
* Patients:
* Additional pathologies that influence the mobility of the ankle joint
* Bilateral surgery
* Use of walking aids
* Healthy control group:
* Lower extremity surgery
* Pain in the lower extremities within the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 patients who had undergone lengthening osteotomy of the lateral column of the foot 2 to 10 years prior and 20 age and sex matched healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Passive plantarflexion and dorsiflexion range of motion | 0 months
  measured using a Biodex

SECONDARY OUTCOMES:
3D hindfoot and forefoot range of motion during level and uphill walking | 0 months
  assessed as max plantarflexion to max dorsiflexion of the ankle using marker and camera based motion capture
Isokinetic strength in plantarflexion, dorsiflexion, inversion, and eversion | 0 months
  Max moment assessed using a Biodex
Lower leg muscle activation | 0 months
  Max electromyographic signal intensity
Clinical outcome | 0 months
  assessed by American Orthopaedic Foot and Ankle Society (AOFAS) Hindfoot Score (questionnaires) (best score: 100 - no limitations)
Functional outcome | 0 months
  assessed by Foot Function Index (questionnaire) (best score: 0; worst score 100)

CONTACTS AND LOCATIONS:
Overall Officials: Corina Nüesch, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No